CLINICAL TRIAL: NCT02773979
Title: A Phase 1 Dose Escalation Trial to Assess the Safety and Efficacy of Infectious (Replication-intact), Cryopreserved Plasmodium Falciparum Sporozoites (PfSPZ Challenge) Administered by Direct Venous Inoculation Under Chloroquine Cover (PfSPZ-CVac) on Varying Schedules in Healthy Malaria-Naïve Adults in the United States
Brief Title: PfSPZ Challenge in Healthy Malaria-Naïve Adults in the United States
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11-0042; HHSN272201300019I
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2017-04-05

CONDITIONS: Plasmodium Falciparum Infection
Keywords: challenge; malaria; P. falciparum; PfSPZ; sporozoites; vaccine
MeSH Terms: conditions — Malaria | interventions — Chloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: PfSPZ 51200 sporozoites/Placebo (Active Comparator): Chloroquine (CQ)/PfSPZ Challenge 51200 sporozoites or CQ/normal saline (NS). N=12, randomized 3:1
  Interventions: Drug: Chloroquine; Biological: PfSPZ (NF54) Challenge; Other: Placebo
- Group 2: PfSPZ 102400 sporozoites/Placebo (Active Comparator): CQ/PfSPZ Challenge 102400 sporozoites or CQ/NS. N=4, randomized 3:1
  Interventions: Drug: Chloroquine; Biological: PfSPZ (NF54) Challenge; Other: Placebo
- Group 3: PfSPZ 102400 sporozoites (Active Comparator): CQ/PfSPZ Challenge 102400 sporozoites N=9
  Interventions: Drug: Chloroquine; Biological: PfSPZ (NF54) Challenge

INTERVENTIONS:
Drug: Chloroquine — Administered as 600mg PO, day 1, 300mg PO days 8, 15, 22.
Biological: PfSPZ (NF54) Challenge — Cryopreserved Plasmodium falciparum (Pf) fully infectious sporozoites (SPZ) that have been developed to be used to infect volunteers in controlled human malaria infection (CHMI) to assess the efficacy of antimalarial drugs and vaccines. The PfSPZ (NF54) Challenge contains a laboratory malaria strain isolated from a Dutch traveler to Africa.
Other: Placebo — Placebo
  Arms: Group 1: PfSPZ 51200 sporozoites/Placebo; Group 2: PfSPZ 102400 sporozoites/Placebo

SUMMARY:
This phase I trial of the replication-intact PfSPZ Challenge vaccine given under CQ cover will enroll 28 healthy volunteers to receive PfSPZ or placebo, as well as suppressive doses of chloroquine (CQ)on varying schedules. 10 weeks post 3rd immunization subjects will be subjected to controlled human malarial infection. The primary objective of this study is to evaluate the safety and tolerability of escalating doses of Sanaria PfSPZ Challenge administered by DVI on varying schedules to healthy malaria-naïve adults taking suppressive doses of CQ (PfSPZ-CVac).

DETAILED DESCRIPTION:
This phase I trial of the replication-intact PfSPZ Challenge vaccine given under CQ (PfSPZ-CVac) cover will randomize 28 healthy adult participants to one of three cohorts. Group 1 (n=12) will be randomized to receive PfSPZ Challenge vaccine at a dose of 51,200 sporozoites or 0.5 mL of sterile normal saline placebo by DVI on Days 3, 10 and 17. Group 2 (n=4) will be randomized to receive PfSPZ Challenge vaccine at a dose of 102,400 sporozoites or 0.5 mL of sterile normal saline placebo by DVI on Days 3, 10, and 17. Within both groups, placebo will be assigned 1:3, with blinded allocation to the two treatments within each group. All subjects in Study Groups 1 and 2 will receive, by directly observed treatment (DOT), oral chloroquine (CQ) on Days 1, 8, 15, and 22 at a suppressive dose of 600 mg base on Day 1 and 300 mg base on Days 8, 15 and 22. All subjects in Group 3 (n=9) will receive PfSPZ Challenge vaccine at a dose of 102,400 sporozoites per administration, with vaccine given on a Day 1, 6, and 11 schedule. Subjects in Group 3 will also receive, by DOT, oral CQ, with a suppressive dose of 600 mg base on Day 1 and a dose of 300 mg base on Days 6, 11, and 16. At 10 weeks after the third administration of study vaccine or placebo, all subjects within the three groups will receive the PfSPZ Challenge by direct venous injection at a dose of 3,200 P. falciparum sporozoites to assess vaccine efficacy against controlled human malarial infection (CHMI). The primary objective of this study is to 1) evaluate the safety and tolerability of escalating doses of Sanaria PfSPZ Challenge administered by DVI on varying schedules to healthy malaria-naïve adults taking suppressive doses of CQ (PfSPZ-CVac).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults (males and non-pregnant, non-lactating females) between the ages of 18 and 45 years, inclusive.
2. Able and willing to participate for the duration of the study.
3. Able and willing to provide written (not proxy) informed consent.
4. Provides informed consent before any study procedures, correctly answers >/= 70% of questions on the post consent quiz and is available for all study visits.
5. Women of childbearing potential* must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to each vaccination and on the day of malaria challenge.

   * Not sterilized via bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or menopausal and still menstruating or < 1 year of the last menses.
6. Women of childbearing potential must have used an acceptable method of contraception* in the 30 days prior to enrollment and must agree to continue use of the same method throughout the study.

   * Includes, but is not limited to, abstinence from sex with men, monogamous relationship with vasectomized partner who has been vasectomized for 6 months or more prior to enrollment, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing, successful Essure placement (permanent, non-surgical, non-hormonal sterilization) with documented confirmation test at least 3 months after the procedure, and licensed hormonal methods such as implants, injectables, or oral contraceptives.
7. Is in good health, as judged by the investigator, and determined by vital signs (heart rate, blood pressure, and oral temperature), medical history and physical examination.
8. Able to understand and comply with planned study procedures.
9. Reachable (24/7) by mobile phone during the whole study period and willing to provide two close contacts to assist with making contact.
10. Lives in the greater Seattle area and within an approximately one hour commute to the study research clinic.
11. Willing to avoid non-study related blood donation for 3 years following P. falciparum challenge.
12. Agrees not to travel to a malaria endemic region during the entire course of the trial.
13. Agrees not to travel away from the greater Seattle area from the day of first study immunization through 20 days after the last study immunization, and during the 29 days after CHMI.

Exclusion Criteria:

1. History of malaria infection or vaccination, residence in a malaria-endemic area for > / =5 years, travel to a malaria-endemic area in the past 6 months, or participation in a malaria research study.
2. Is breastfeeding or plans to breastfeed at any time throughout the study.
3. Plans to become pregnant at any time throughout the study.
4. Use of any antimalarial antibiotic or drug within 28 days prior to Study Day 1 or planned use during the study period.
5. Any clinically significant acute or chronic medical condition* or need for chronic medications** that, in the opinion of the investigator, will interfere with immunity or affect safety.

   * Includes, but is not limited to, disorders of the liver, kidney, lung, heart, or nervous system, or other metabolic or autoimmune/inflammatory conditions.

     * Receipt of systemic, prescription medications for the treatment of chronic medical conditions or variations of normal physiologic functions are permissible if, in the opinion of the investigator, they are used for conditions that are not clinically significant and would not impact the effectiveness of the vaccine or the safety of the subject or the safety and immunogenicity outcomes of the protocol. Use of systemic, over-the-counter medications and PRN systemic, prescription medications are allowed if, in the opinion of the investigator, they pose no additional risk to subject safety, vaccine efficacy or assessment of immunogenicity/reactogenicity. Topical (except corticosteroid) medications, nasal (including corticosteroid) medications, vitamins, and supplements are permissible. Any drug with antimalarial properties is not permissible.
6. Asthma, other than mild, well-controlled asthma*.

   * Cold or exercise induced asthma controlled with inhaled medications other than inhaled corticosteroids is permissible. Subjects should be excluded if they require daily bronchodilator use, or have had an asthma exacerbation requiring oral/parenteral steroid use or have used theophylline or inhaled corticosteroids in the past year.
7. Diabetes mellitus.
8. History of a psychiatric condition that may make study compliance difficult, such as schizophrenia, or unstable bipolar disorder*.

   * Includes persons with psychoses or history of suicide attempt or gesture in the 3 years before study entry or an ongoing risk for suicide.
9. Any history of non-febrile seizures or complex febrile seizures*

   * History of simple febrile seizures or a family history of seizure disorder is not exclusionary
10. Autoimmune disease (autoimmune thyroid disease is permissible and vitiligo or mild eczema not requiring chronic therapy is permissible).
11. Known or suspected congenital or acquired immunodeficiency including anatomic or functional asplenia* or immunosuppression as a result of underlying illness or treatment. *Any splenectomy is exclusionary.
12. Abuse of alcohol or drugs that, in the opinion of the investigator, may interfere with the subject's ability to comply with the protocol.
13. Body mass index (BMI) > / = 35 kg/m^2.
14. Active neoplastic disease*.

    * Subjects with a history of malignancy may be included if treated by surgical excision or if treated by chemotherapy or radiation therapy and has been observed for a period that in the investigator's estimation provides a reasonable assurance of sustained cure (not less than 36 months).
15. Chronic topical or systemic corticosteroid use*.

    * Corticosteroid nasal sprays for allergic rhinitis are permissible. Persons using a topical corticosteroid for a limited duration for mild uncomplicated dermatitis such as poison ivy or contact dermatitis may be enrolled the day after their therapy is completed. Oral or parenteral (IV, SC, or IM) corticosteroids given for non-chronic conditions not expected to recur are permissible if, within the year prior to enrollment, the longest course of therapy was no more than 14 days and no oral or parenteral corticosteroids were given within 30 days prior to enrollment. Intraarticular, bursal, tendon, or epidural injections of corticosteroids are permissible if the most recent injection was at least 30 days prior to enrollment.
16. Receipt or planned receipt of inactivated vaccine or allergy desensitization injection from 14 days before the first immunization through 14 days after the last immunization.
17. Planned receipt of inactivated vaccine or allergy desensitization injection from 14 days prior to CHMI through 28 days after CHMI.
18. Receipt or planned receipt of live attenuated vaccine 30 days before or at any time during the study up to 28 days after CHMI.
19. Receipt of any experimental agent* within 30 days prior to enrollment or planned receipt prior to the end of the study.

    * Vaccine, drug, biologic, device, blood product, or medication.
20. Plans to enroll in another clinical trial* that could interfere with safety assessment of the investigational product at any time during the study period.

    * Includes trials that have a study intervention such as a drug, biologic, or device.
21. Receipt of blood products or immunoglobulin within six months prior to Study Day 1 or donation of a unit of blood within two months before Study Day 1.
22. Systolic blood pressure > / = 161 mm Hg or diastolic blood pressure > / = 96 mm Hg.
23. Resting heart rate < 55 or > 100 beats per minute.
24. Oral temperature > / = 38 degrees C (100.4 degrees F).
25. Positive serology for HIV 1/2.
26. Positive hepatitis B surface antigen (HBsAg).
27. Positive antibody to hepatitis C virus (HCV).
28. Any Grade 1 or higher screening clinical lab value* (see Toxicity Tables Section 9.2.3).

    * Screening clinical labs include blood tests (white blood cells [WBC], hemoglobin, platelets, creatinine, non-fasting glucose, potassium, alanine aminotransferase [ALT], aspartate aminotransferase [AST], alkaline phosphatase, and total bilirubin) and urine dipstick tests (protein, glucose, hemoglobin). Any Grade 1 or higher value for any screening test will exclude the subject from enrollment with the exception of hematuria > / = 1 + detected during menses or other endometrial bleeding for females. In this situation, the test can be repeated if clinically warranted but is not considered an indicator of poor health status or increased risk and so is not a contraindication to enrollment.
29. Acute febrile illness (oral temperature > / = 38 degrees C [100.4 degrees F]) or other acute illness within 3 days prior to vaccination (subject may be rescheduled).
30. A screening ECG with abnormalities consistent with underlying heart disease.*

    * Pathologic Q waves and significant ST-T wave changes; left ventricular hypertrophy; any non-sinus rhythm excluding isolated premature atrial or ventricular contractions; right or left bundle branch block; QT/QTc interval > 450 ms; or advanced (secondary or tertiary) A-V heart block.
31. Has a history of psoriasis or porphyria.
32. Has a known allergy to chloroquine, 4-aminoquinoline derivatives, atovaquone, proguanil,artemether-lumenfantrine, 8-aminoquinoline derivatives, non-steroidal anti- inflammatory drugs, or acetaminophen.
33. Is using or intends to use a medication that is cross-reactive with CQ** or atovaquone and proguanil, such as cimetidine or metoclopramide, during the study period.

    * Antacids and kaolin can be administered at least 4 hours from intake of chloroquine.

      * Does not apply to infectivity controls
34. History of retinal or visual field changes, clinically significant auditory damage, or G6PD deficiency.
35. Has history of or a positive test for sickle cell disease or trait or other hemoglobinopathy.
36. Plans to undergo surgery (elective or otherwise) between enrollment and the end of the study.
37. Known hypersensitivity to PfSPZ or its components.
38. Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
The number of serious adverse events (SAEs) related to study product. | Days 1-203
The number of solicited local adverse events (AEs) | Days 1-93
The number of solicited systemic adverse events(AEs) | Day 1-116
The number of unsolicited adverse events (AEs) related to study product | Days 1-130
The severity of solicited local adverse events (AEs) as assessed by grading scales | Day 1-93
The severity of solicited systemic adverse event (AEs) as assessed by grading scales | Day 1-116
The severity of unsolicited AEs related to study product as assessed by grading scales. | Days 1-130

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Washington Health Research Institute - Vaccines and Infectious Diseases, Seattle, Washington, United States

REFERENCES:
- [Derived] Murphy SC, Deye GA, Sim BKL, Galbiati S, Kennedy JK, Cohen KW, Chakravarty S, Kc N, Abebe Y, James ER, Kublin JG, Hoffman SL, Richie TL, Jackson LA. PfSPZ-CVac efficacy against malaria increases from 0% to 75% when administered in the absence of erythrocyte stage parasitemia: A randomized, placebo-controlled trial with controlled human malaria infection. PLoS Pathog. 2021 May 28;17(5):e1009594. doi: 10.1371/journal.ppat.1009594. eCollection 2021 May. PMID 34048504